CLINICAL TRIAL: NCT00302276
Title: Weight Loss Maintenance of a New Bioactive Compound (Metobes-Long)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KF11-150/03
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-11

CONDITIONS: Obesity
Keywords: Body fat loss; energy expenditure; capsaicin; caffeine; green tea; calcium; fecal fat; fecal energy
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Drug: Metobes-compound

SUMMARY:
The objective of the present study was to investigate the acute and sub-chronic effect of a supplement containing green tea extract, capsaisin, caffeine, tyrosine and calcium or placebo taken t.i.d on thermogenesis, body fat loss, and fecal fat excretion. Furthermore, if a 8-week supplementation could prevent weight-regain after initial 4-week weight loss.

DETAILED DESCRIPTION:
It has previously been shown that a combination of tyrosine, capsaicin, catechines, and caffeine may stimulate the sympathetic nervous system and promote satiety, lipolysis and thermogenesis. In addition, dietary calcium may increase fecal fat excretion.

Method:

80 healthy Danish overweight to obese (BMI between 28 and 35 kg/m2), 18 to 70 years of age subjects of both gender. All subjects was be weight stable (within 3-kg) 2 months prior to study inclusion, non-smoking, non-athletic and have no daily use of medication except for anticonception and antihypertensive compounds. All subjects gave their written consent after verbal and written information about the study. The study protocol was approved by The Municipal Ethical Committee of Copenhagen and Frederiksberg as being in accordance with the Helsinki II Declaration.

The total study period was 12 weeks. The intervention design was an 8-weeks randomized, 3-arm parallel, placebo-controlled and double-blind intervention. Prior to the randomized intervention a weight loss was initiated by 4 week treatment on a 3.4 MJ/d low caloric diet (LCD). Only subject who lost more than 4% of their initial body weight after 4 weeks LCD treatment was randomized and continued in the study.

The subjects were randomized into 3 balanced groups i.e. placebo, simple or enterocoated release. All subjects received dietary instruction to a slightly hypo caloric diet of -300 kcal/day after the isoenergetic educational system. The dietary advice was reinforced by dietetic consultations every fortnight.

Body weight and composition were assessed by DEXA before and after the LCD period, four weeks into the randomized period and at completion i.e. the last day of the study.

All participants underwent assessment of energy expenditure by indirect calorimetry in a ventilated hood. The first respiratory measurement was on the first day of the intervention and will last for 5 hours.

All subjects collected all feces excreted three days prior to respiratory measurement and one day of urine excreted.

ELIGIBILITY:
Inclusion Criteria:

* healthy Danish overweight to obese (BMI between 28 and 35 kg/m2), 18 to 70 years of age subjects of both gender. All subjects must be weight stable (within 3-kg) 2 months prior to study inclusion.

Exclusion Criteria:

* smokers, athletic, daily use of medication except for anticonception and antihypertensive compounds, blood pressure above 165/95 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-01; Study Completion 2004-07

PRIMARY OUTCOMES:
Body weight, fat mass, fat free mass, energy expenditure, respiratory quotient, fecal fat, fecal energy

SECONDARY OUTCOMES:
blood pressure, heart rate, urine catecholamines, self-reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kondrup, Prof, Principal Investigator — Department of Human Nutrition, The Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark